CLINICAL TRIAL: NCT04837859
Title: Phase II Trial of Individualized Immunotherapy in Early-Stage Unfavorable Classical Hodgkin Lymphoma
Acronym: INDIE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Paul Broeckelmann, Priv. Doz., University of Cologne
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-4470
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A age 18-60 (Experimental): Patients at the age of 18-60 years at enrollment will receive 2 initial doses of 200 mg tislelizumab in 21-day intervals followed by an interim positron emission tomography (PET-2). Following a PET-guided approach, patients with a negative PET-2 (i.e. Deauville score 1-3) according to central review will continue receiving tislelizumab for another 4 doses of 300 mg in 28-day intervals. Patients with a positive PET-2 (i.e. Deauville score >3) will receive 4 cycles of combined 300 mg tislelizumab on day 1 and AVD chemotherapy on day 1 and 15 in 28-day cycles (4x T-AVD). For all patients, 30 Gy involved-site radiotherapy (IS-RT) will only be applied in case of PET positivity after completion of (chemo-) immunotherapy.
  Interventions: Drug: Tislelizumab
- Arm B Age 60+ (Experimental): Patients above the age of 60 years will be enrolled in a separate, exploratory cohort and receive PET-guided treatment with tislelizumab or T-AVD as described above. However, all patients in the exploratory cohort for older patients will receive consolidating 30 Gy IS-RT.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — age 18-60: Tislelizumab alone or in combination with AVD (depending on the PET result after 2x Tislelizumab) followed by IS-RT if PET positive resudues after the end of Tis or Tis-AVD age 60+: Tislelizumab alone or in combination with AVD (depending on the PET result after 2x Tislelizumab) followed by IS-RT for all patients

SUMMARY:
The aim of the trial is to establish an individualized first-line treatment incorporating checkpoint inhibition for early-stage unfavorable cHL, which is effective and well tolerated.

DETAILED DESCRIPTION:
Programmed cell death protein-1 (PD-1) blockade is highly effective and well tolerated in relapsed or refractory cHL and has also demonstrated efficacy in the first-line treatment of cHL in combination with doxorubicin, vinblastine, and dacarbazine (AVD) in the phase II GHSG NIVAHL trial. A relevant proportion of patients achieved an early metabolic complete remission (CR) with anti-PD-1 monotherapy and might not require standard chemo- or radiotherapy. Limiting therapy-associated short- and long-term side effects of these conventional treatments including impaired quality of life, second primary malignancies or organ damage is of utmost importance in the predominantly young cHL patients. This trial will hence further reduce treatment intensity and provide a chemo- and radiotherapy-free therapy to optimally responding patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 for the main trial cohort
* Age ≥ 61 years and eligible for AVD as determined by CIRS-G score and investigator for the exploratory cohort
* First diagnosis of treatment-naïve cHL
* Early-stage unfavorable disease (i.e. stage IA, IB and IIA with risk factors a-d, stage IIB with risk factors c-d):

  1. large mediastinal mass
  2. extranodal lesion(s)
  3. elevated erythrocyte sedimentation rate
  4. ≥ 3 nodal areas

     Exclusion Criteria:
* Presence of nodular-lymphocyte predominant Hodgkin lymphoma, grey-zone lymphoma and/or central nervous system involvement of lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paul Broeckelmann, Dr., Principal Investigator — 1st Department of Medicine, Cologne Universit Hospital
Locations (1):
- 1st Department of Medicine, Cologne University Hospital, Cologne, Germany